CLINICAL TRIAL: NCT02832115
Title: Topical Nitroglycerine Treatment for Radial Artery Spasm Prevention
Acronym: TNT-RASP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Principal Investigator, Prabhakaran Gopalakrishnan, Prabhakaran Gopalakrishnan, MD, Aultman Health Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016.04.PG
Record Dates: First submitted 2016-06-26; First posted 2016-07-14 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Radial Artery Spasm; Angina; Coronary Artery Disease
Keywords: Cardiac Catheterization; Vascular Access Site Complications; Vasodilator; Nitroglycerine; Lidocaine
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease | interventions — Nitroglycerin; Vasodilation; Lidocaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study (Experimental): 40 mg of topical lidocaine and 30 mg of topical nitroglycerine is applied to the wrist overlying radial pulse (centered approximately 1 inch proximal to the radial styloid process) at least 60 minutes before arterial puncture. Immediately prior to sterile preparation of access site, transdermal preparation will be removed in the cath lab.
  Interventions: Drug: Topical Nitroglycerine; Drug: Topical Lidocaine
- Control (Placebo Comparator): 40 mg of topical lidocaine and placebo is applied to the wrist overlying radial pulse (centered approximately 1 inch proximal to the radial styloid process) at least 60 minutes before arterial puncture. Immediately prior to sterile preparation of access site, transdermal preparation will be removed in the cath lab.
  Interventions: Drug: Topical Lidocaine

INTERVENTIONS:
Drug: Topical Nitroglycerine — Topical nitroglycerine is applied to wrist prior to transradial cardiac catheterization to dilate radial artery and reduce spasm in study arm patients
  Other Names: Vasodilation
  Arms: Study
Drug: Topical Lidocaine — Topical Lidocaine is applied to wrist prior to transradial cardiac catheterization in both study and control arms
  Other Names: Topical anesthetic

SUMMARY:
The primary objective of the study is to determine the role of transdermal vasodilators as an adjunct to parenteral vasodilators in reducing radial artery spasm, improving patient comfort, and post procedure radial artery patency during transradial coronary angiograms and interventions. The study hypothesis is that transdermal vasodilators will increase radial artery size and reduce radial artery spasm as well as improve patient comfort and post procedure radial artery patency. This is a single-center, double-blind, randomized, placebo-controlled study comparing the effect of transdermal preparations of lidocaine + nitroglycerine and lidocaine + placebo on radial artery spasm in patients undergoing transdermal coronary angiograms. Prior to the procedure, each patient will be randomized into either the control arm, lidocaine + placebo, or study arm, lidocaine + nitroglycerine.

DETAILED DESCRIPTION:
Background:

Vascular access site complications (VASC) during cardiac catheterizations are significantly higher in femoral access compared to radial access. Main disadvantage in radial access is the restriction in size of catheters as well as incidence of radial artery spasm. Radial spasm is identified by pain in the forearm aggravated by movement of the catheter/sheath; difficulty in manipulating the catheter; loss of radial pulse or damping of radial arterial pressure. Tortuosity and loops in upper extremity arterial tree could mimic some findings of radial artery spasm. Incidence of radial spasm has been reported to range between 4% and 20%. Risk factors include smaller radial artery diameter, atherosclerotic lesions, entrance of guidewires into side branches, vessel tortuosity, larger arterial sheath diameters, procedure duration, female sex, younger age, lower BMI, Diabetes, number of catheters used, volume of contrast, unsuccessful access at first attempt, fear and anxiety. Mean size of radial artery is reported at 2.44 mm. Women and persons of south Asian descent tend to have smaller radial arteries with means of 1.91mm and 2.00 mm respectively. Outer diameters of commonly used 5 French (5F) and 6 French (6F) sheaths are 2.16 mm and 2.62 mm respectively. Ratio of radial artery to sheath size affects post-procedural radial artery flow.

Transdermal vasodilators prior to vascular access would increase chance for successful arterial access in first attempt and increase radial artery to sheath size ratio both of which should have additive benefit to intraarterial (IA) vasodilators in reducing spasm. Transdermal lidocaine would reduce pain during subcutaneous lidocaine, which can further ameliorate the risk of radial artery spasm. Use of transdermal nitroglycerine has been shown to safely increase radial artery size without significant hypotension.

Aim:

To study the role of transdermal vasodilators as an adjunct to parenteral vasodilators, in reducing radial artery spasm and improving patient comfort and post procedure radial artery patency during radial coronary angiograms and interventions.

Hypothesis:

Transdermal vasodilators will increase radial artery size and reduce radial artery spasm as well as improve patient comfort and post procedure radial artery patency.

Study Design:

Single center, double blinded, randomized placebo-controlled study comparing effect of transdermal preparations of lidocaine + Nitroglycerine and lidocaine + placebo on radial artery spasm and procedural success in patients undergoing radial coronary angiograms and interventions. All patients will receive standard parenteral cocktail including intraarterial or intravenous (IV) heparin and IA nitroglycerine and / or verapamil. Exact doses and combinations would be at the discretion of individual provider based on patient's hemodynamic status and comorbid conditions.

End Points:

Primary:

1. Radial artery spasm: Incidence of radial artery spasm indicated by a Radial artery spasm score of 1 or more. Radial artery spasm score is sum of:

a. Verbal or nonverbal expression of discomfort in the forearm during catheter/sheath manipulation - Absent :0; Present:1 b. Difficulty in manipulating the catheter- Absence :0; Present:1 c. Difficulty with sheath removal: Absent: 0; Present:1 d. Additional use of IA nitroglycerine or verapamil after the initial vasodilator cocktail for suspected radial artery spasm- No:0; Yes:1.

Secondary:

1. Change in ipsilateral radial artery dimension (mm) before application of topical nitroglycerine / placebo (pre-dilation) vs. prior to arterial puncture after application of topical nitroglycerine / placebo (Post-dilation).
2. Procedural failure: Need to abort procedure or convert to femoral approach.
3. Patient forearm discomfort or pain during procedure measured using Visual analog scale 0-10.
4. Ipsilateral radial pulse at end of procedure 0-4+.

Safety endpoints:

1. Asymptomatic Hypotension: Systolic blood pressure (SBP) < 90 mm Hg
2. Symptomatic Hypotension: Dizziness or lightheadedness and SBP < 100 mm Hg
3. Intractable headache unrelieved by 1gm of acetaminophen

Adverse Effects of investigational product:

1. Hypotension: SBP < 90 mm Hg requiring intervention any time after application of investigational product (IP) in Ambulatory Cardiac Unit (Same Day) until removal of IP in cathlab
2. Dizziness or lightheadedness requiring intervention any time after application of IP in Ambulatory Cardiac Unit (Same Day) until removal of IP in cathlab
3. Headache requiring intervention anytime after application of IP in Ambulatory Cardiac Unit (Same Day) until removal of IP in cathlab

Complications of Radial artery catheterization:

1. Forearm hematoma > 5cm 2. Absent ipsilateral radial pulse (0) after procedure

Methods:

1. Patient enrollment:

   a. Outpatient: i. Whenever feasible, information about the study would be provided to the patient prior to arrival in Ambulatory Cardiac Unit (Same Day) (preferably at the time of scheduling). When not feasible, patients will be contacted via phone prior to the day of procedure or approached in the Ambulatory Cardiac Unit (Same Day) unit on the day of the procedure by one of the investigators to assess interest in participation.

   ii. Patients who are interested and meet all inclusion criteria and none of the exclusion criteria will be enrolled in the trial in the Ambulatory Cardiac Unit (Same Day) on the day of their scheduled procedure. One of the participating investigators will obtain informed consent after the patient has had time to review the consent and all questions have been answered.

   b. Inpatient: i. Hospitalized patients who are interested and meet all inclusion criteria and none of the exclusion criteria may be enrolled in the trial on or before the day of their scheduled procedure, but always prior to transfer to the Catheterization Lab. One of the participating investigators will obtain informed consent after the patient has had time to review the consent and all questions have been answered.
2. After reviewing the most current vital signs, patients without any exclusion criteria will be randomized 1:1 to control arm (40 mg Lidocaine + placebo) or study arm (40 mg lidocaine + 30 mg nitroglycerine)
3. Study drug assignment will be randomized and distributed by a delegated member of the study staff, with oversight by the PI or Sub-Is, for patients consented and enrolled in the trial at least 60 minutes prior to the procedure start time.
4. Pre-medication cross sectional image of ipsilateral radial artery (approximately 1 inch proximal to radial styloid process) will be recorded using bedside sonogram with no more than gentle pressure and site marked with a skin marker.
5. Ipsilateral wrist circumference (1 inch proximal to radial styloid process) will be documented.
6. Pre-procedure ipsilateral radial pulse strength (0-4+) will be documented. (4+ Bounding, 3+ Increased, 2+ Normal, 1+ Weak, 0+ Absent or nonpalpable)
7. Transdermal preparation will be applied to ipsilateral wrist overlying radial pulse (centered approximately 1 inch proximal to radial styloid process) at least 60 minutes before procedure start time at a dose of 40mg (6 ribbons of 2 inches each) of 5% Lidocaine and 30mg (8 ribbons of 2 inches each) of 2% Nitroglycerine/Placebo.
8. Patients will complete the Amsterdam Preoperative Anxiety and Information Scale (APAIS).
9. Vitals signs to be checked every 30 minutes (±10 minutes) after application of the topical preparation for 60 minutes (±10 minutes) then every 60 minutes (±10 minutes) until procedure.
10. If SBP < 100 mm Hg and patient complains of dizziness or light-headedness or if SBP < 90 mm Hg, the topical preparation will be removed promptly, 250 ml of 0.9% Normal Saline (NS) IV bolus will be given over 15 minutes, and provider will be notified immediately.
11. If patient complains of headache, one or two tablets of 500 mg acetaminophen will be given by mouth every 4 hours as needed. One tablet will be given if the patient reports a value of 0-3 on the pain scale, and two tablets will be given if the patient reports a value of 4 or greater on the pain scale. The maximum dose of acetaminophen is 4g in 24 hours.
12. If 30 minutes after acetaminophen administration, headache intensity ≥ 5/10 or patient unable to tolerate intensity of headache, the topical preparation will be removed promptly and provider will be notified immediately.
13. If any of the safety endpoints occur, an investigator will be notified immediately and further decision to proceed with cardiac catheterization or additional workup or treatment would be at the discretion of the investigator.
14. Immediately prior to sterile preparation of access site, transdermal preparation will be removed in Cath Lab and post-dilation cross sectional image of ipsilateral radial artery (approximately 1 inch proximal to radial styloid process) will be captured using bedside sonogram applying no more than gentle pressure.
15. Conscious sedation with IV fentanyl and midazolam given with exact dosing at operator's discretion (based on patient's hemodynamic status and comorbid conditions).
16. After sterile preparation 0.5 - 1.0 ml of subcutaneous lidocaine is administered and radial artery cannulated using modified seldinger technique with 5F or 6F hydrophilic sheath.
17. Parenteral radial cocktail (IV/IA heparin +/- IA nitroglycerine +/- IA verapamil) is given with exact combination and dose at discretion of operator based on patient's hemodynamic status.
18. Coronary angiogram and or intervention performed adopting best practices with care to minimize procedure time, contrast volume and catheter exchanges and avoiding side branches.
19. Following parameters are documented:

    1. Patient demographics (Age, Sex, BMI, Race)
    2. Conscious sedation drugs and doses used
    3. Sheath size
    4. Number of arterial sticks before arterial access: One or more (Blood in arteriotomy needle equates arterial stick)
    5. Wire passage in one or more attempts
    6. Sheath insertion in one or more attempts
    7. Radial parenteral cocktail used
    8. Radial artery spasm score:
    9. Verbal or nonverbal expression of discomfort in the forearm during catheter/sheath manipulation - Absent:0; Present:1 ii. Difficulty in manipulating the catheter - Absent:0; Present:1 iii. Difficulty in sheath removal - Absent:0; Present:1 iv. Additional use of IA nitroglycerine or verapamil after the initial vasodilator cocktail for suspected radial artery spasm - No:0; Yes:1

    i. Use of long sheath j. Use of hydrophilic wires or catheters k. Tortuosity of upper extremity vessels / anatomic variants l. Catheters used m. Contrast volume n. Difficulty in removing catheters and sheath o. Use of IA/IV nitroglycerine and/or verapamil at end of procedure for sheath removal: provisional use when radial artery spasm present or suspected vs. routine pre-emptive use to avoid radial artery spasm per operator standard practice.

    p. Length of procedure q. Change to femoral arterial access and reason r. Procedures performed
20. Patient's perceived peri-procedure forearm discomfort documented using VAS (1-10) at the completion of the procedure
21. Post procedure strength of ipsilateral radial pulse (0-4+) after radial band removal documented and presence and size of hematoma at access site at time of radial band removal documented
22. For patients who have the sheath left in place for percutaneous coronary intervention (PCI) as a separate procedure at a later time, data will be collected for the initial diagnostic catheterization only. The procedure will be considered completed with removal of last diagnostic catheter. Post procedure pulse will be the radial pulse after the PCI.
23. Patients are monitored for adverse events for the following duration:

    a. For patients discharged home from the ambulatory cardiac unit (same day unit) after procedure completion: i. Until discharged home b. For hospitalized patients: i. Until 120 minutes after Radial band, or comparable product, removal

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Radial artery catheterization

Exclusion Criteria:

1. Hypersensitivity or contraindication to lidocaine
2. Hypersensitivity or contraindication to nitroglycerine
3. Recent use of phosphodiesterase 5 inhibitors (<24 hours after sildenafil or vardenafil; <48 hours after tadalafil)
4. Baseline weak radial pulse (0 or 1+)
5. Baseline hypotension SBP < 100 mmHg at the time of enrollment
6. Dizziness or light-headedness at the time of enrollment
7. Severe Aortic Stenosis or Hypertrophic obstructive cardiomyopathy
8. Previous unknown bypass grafts or known left internal mammary graft
9. Chest pain within 6 hours of IP administration
10. More than 2 episodes of chest pain within 24 hours prior to IP administration
11. Use of sublingual, transdermal, or intravenous nitroglycerine within 6 hours prior to IP administration
12. Likely need for use of nitroglycerine for non-study indication
13. Narcotic or sedative within 4 hours of enrollment
14. Women who are suspected or known to be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prabhakaran Gopalakrishnan, MD, Principal Investigator — Aultman Hospital
Locations (1):
- Aultman Hospital, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siudak Z, Zawislak B, Dziewierz A, Rakowski T, Jakala J, Bartus S, Noworolnik B, Zasada W, Dubiel JS, Dudek D. Transradial approach in patients with ST-elevation myocardial infarction treated with abciximab results in fewer bleeding complications: data from EUROTRANSFER registry. Coron Artery Dis. 2010 Aug;21(5):292-7. doi: 10.1097/MCA.0b013e32833aa6d1. PMID 20453640
- [Background] Hildick-Smith DJ, Walsh JT, Lowe MD, Shapiro LM, Petch MC. Transradial coronary angiography in patients with contraindications to the femoral approach: an analysis of 500 cases. Catheter Cardiovasc Interv. 2004 Jan;61(1):60-6. doi: 10.1002/ccd.10708. PMID 14696161
- [Background] Azzalini L, Tosin K, Chabot-Blanchet M, Avram R, Ly HQ, Gaudet B, Gallo R, Doucet S, Tanguay JF, Ibrahim R, Gregoire JC, Crepeau J, Bonan R, de Guise P, Nosair M, Dorval JF, Gosselin G, L'Allier PL, Guertin MC, Asgar AW, Jolicoeur EM. The Benefits Conferred by Radial Access for Cardiac Catheterization Are Offset by a Paradoxical Increase in the Rate of Vascular Access Site Complications With Femoral Access: The Campeau Radial Paradox. JACC Cardiovasc Interv. 2015 Dec 21;8(14):1854-64. doi: 10.1016/j.jcin.2015.07.029. Epub 2015 Nov 18. PMID 26604063
- [Background] Ho HH, Jafary FH, Ong PJ. Radial artery spasm during transradial cardiac catheterization and percutaneous coronary intervention: incidence, predisposing factors, prevention, and management. Cardiovasc Revasc Med. 2012 May-Jun;13(3):193-5. doi: 10.1016/j.carrev.2011.11.003. Epub 2012 Jan 5. PMID 22226169
- [Background] Saito S, Ikei H, Hosokawa G, Tanaka S. Influence of the ratio between radial artery inner diameter and sheath outer diameter on radial artery flow after transradial coronary intervention. Catheter Cardiovasc Interv. 1999 Feb;46(2):173-8. doi: 10.1002/(SICI)1522-726X(199902)46:23.0.CO;2-4. PMID 10348538
- [Background] Ercan S, Unal A, Altunbas G, Kaya H, Davutoglu V, Yuce M, Ozer O. Anxiety score as a risk factor for radial artery vasospasm during radial interventions: a pilot study. Angiology. 2014 Jan;65(1):67-70. doi: 10.1177/0003319713488931. Epub 2013 May 8. PMID 23657175
- [Background] Kotowycz MA, Johnston KW, Ivanov J, Asif N, Almoghairi AM, Choudhury A, Nagy CD, Sibbald M, Chan W, Seidelin PH, Barolet AW, Overgaard CB, Dzavik V. Predictors of radial artery size in patients undergoing cardiac catheterization: insights from the Good Radial Artery Size Prediction (GRASP) study. Can J Cardiol. 2014 Feb;30(2):211-6. doi: 10.1016/j.cjca.2013.11.021. Epub 2013 Nov 23. PMID 24461923
- [Background] Frangosa C, & Nobleb S. How to transform you into a radialist: tips and tricks. Cardiovascular Medicine 14.10 (2011): 315-24.
- [Background] Majure DT, Hallaux M, Yeghiazarians Y, Boyle AJ. Topical nitroglycerin and lidocaine locally vasodilate the radial artery without affecting systemic blood pressure: a dose-finding phase I study. J Crit Care. 2012 Oct;27(5):532.e9-13. doi: 10.1016/j.jcrc.2012.04.019. Epub 2012 Jun 12. PMID 22699036
- [Background] Beyer AT, Ng R, Singh A, Zimmet J, Shunk K, Yeghiazarians Y, Ports TA, Boyle AJ. Topical nitroglycerin and lidocaine to dilate the radial artery prior to transradial cardiac catheterization: a randomized, placebo-controlled, double-blind clinical trial: the PRE-DILATE Study. Int J Cardiol. 2013 Oct 3;168(3):2575-8. doi: 10.1016/j.ijcard.2013.03.048. Epub 2013 Apr 10. PMID 23582415
- [Background] Yoshizaki T, Tabuchi N, Toyama M. Verapamil and nitroglycerin improves the patency rate of radial artery grafts. Asian Cardiovasc Thorac Ann. 2008 Oct;16(5):396-400. doi: 10.1177/021849230801600511. PMID 18812349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study | Control
Started | 48 | 52
Completed | 48 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.45833333 (9.828223218) | 66.40384615 (9.282620521) | 66.91 (9.466884387)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 27 | 36 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Radial artery Dimension [Mean (Standard Deviation); unit: mm^2] — Radial artery dimension (Cross sectional area) in mm2 before application of study or control drug (Pre-Dilation) Population: Only 87 of the participants had radial artery dimension change measured
  mm^2
    number analyzed (Participants) | 42 | 45 | 87
    (all) | 5.6 (2.221596993) | 6.5 (2.450302073) | 6.1 (2.387930965)

OUTCOME MEASURES:

1. Primary Outcome: Radial Artery Spasm
Description: Incidence of radial artery spasm indicated by a Radial artery spasm score of 1 or more. Radial artery spasm score is sum of:
  1. Intraprocedural pain in the forearm aggravated by movement of the catheter/sheath - Absent :0; Present:1
  2. Difficulty in manipulating the catheter- Absence :0; Present:1
  3. Difficulty with sheath removal: Absent: 0; Present:1
  4. Additional use of intraarterial nitroglycerine or verapamil after the initial vasodilator cocktail- No:0; Yes:1
Time Frame: Intraprocedural: From procedure start to application of radial band. Approximate time 30 to 90 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 48 | 52
Participants | 8 | 15

2. Secondary Outcome: Change in Radial Artery Dimension Measured in mm^2.
Description: Change in Radial artery cross sectional area in mm^2 - Before application of topical nitroglycerine / placebo (Pre dilation) vs Prior to arterial puncture after application of topical nitroglycerine / placebo (Post-dilation)
Time Frame: Application of nitroglycerine / placebo until prior to arterial puncture. Approximate 60 to 120 minutes
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Study | Control
Number analyzed (Participants) | 42 | 45
mm^2 | 2.5 (1.668937229) | -0.2 (1.060927244)

3. Secondary Outcome: Number of Patients With Procedural Failure
Description: Need to abort procedure or convert to transfemoral access
Time Frame: Intraprocedural: From procedure start to application of radial band. Approximate time 30 to 90 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 48 | 52
Participants | 0 | 4

4. Secondary Outcome: Patient Discomfort or Pain During Procedure (Visual Analog Scale 0-10)
Description: Patient discomfort or pain during procedure measured using Visual analog scale 0-10, 0 being no discomfort or pain (best) and 10 being worst discomfort or pain (worst)
Time Frame: Intraprocedural: From procedure start to application of radial band. Approximate time 30 to 90 minutes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study | Control
Number analyzed (Participants) | 48 | 48
score on a scale | 0.792 (2.030582155) | 0.875 (1.964529206)

5. Secondary Outcome: Radial Pulse at End of Procedure
Description: Radial pulse at end of procedure 0- 4+, 0 indicating no palpable pulse (worst); 1 + indicating a faint, but detectable pulse; 2 + suggesting a slightly more diminished pulse than normal; 3 + is a normal pulse; and 4 + indicating a bounding pulse (best).
Time Frame: At the end of transradial cardiac catheterization after sheath removal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study | Control
Number analyzed (Participants) | 48 | 48
score on a scale | 2.208333333 (0.650967638) | 2.166666667 (0.558620388)

ADVERSE EVENTS:
Time Frame: Duration of Hospitalization during index procedure: 6 to 48 hours. Typically less than 8 hours if no intervention.
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 5/48 | 5/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study (N=48) | Control (N=52)
Headache (General disorders) | 2 (2) | 1 (1) — Headache reported or requiring Tylenol use
Hematoma < 5 cm (Vascular disorders) | 3 (3) | 4 (4) — Hematoma at Radial access site or Femoral hematoma

LIMITATIONS AND CAVEATS:
Slow enrollment leading to smaller sample than initially planned (100 instead of 150) Radial artery dimensions available in only 87 out of 100 participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT02832115/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-10-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT02832115/Prot_SAP_001.pdf